CLINICAL TRIAL: NCT04348955
Title: Interest of Touch-massage in Hospital Day Care
Acronym: TOMAS
Status: Completed | Type: Observational
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Other Study IDs: ICO-2019-08
Record Dates: First submitted 2020-03-25; First posted 2020-04-16 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Breast Neoplasm Malignant Female
Keywords: Breast cancer; Touch massage; anxiety; chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- women with adjuvant breast cancer: Women between 18 and 70 years old with an adjuvant breast cancer histologically characterized
  Interventions: Behavioral: Women between 18 and 70 years old with an adjuvant breast cancer histologically characterized

INTERVENTIONS:
Behavioral: Women between 18 and 70 years old with an adjuvant breast cancer histologically characterized — Quality of life and anxiety questionnaires before the course of chemotherapy (C1 and C4).
  Touch-Massage during the course of chemotherapy (from C1 to C3) Anxiety questionnaire at the end of the course of chemotherapy (from C1 to C3)

SUMMARY:
In spite of progresses made in the medical and nurse announcement (linked to the cancer plan), still a lot of patients fell lost, anxious, especially during the first venue at the hospital day care for their chemotherapy. A longer time is necessary to give them again explanation, to reassure and to listen to them. However, patients are not always in ability to hear due to their psychological status. Young women seem to be more in distress, this is linked to the fear of the disease, the change of their social status and the future of their children.

It must be noted that there is an increase of complementary therapies including Touch-Massage. Studies showed its interest on quality of life, anxiety, pain and fatigue.

The concept Touch-massage (TM) is defined as a benevolent concern that takes shape through the touch and the sequence of gesture on all or parts of the body. This allows to calm, to relax, to get back into shape, to reassure, to communicate or simply to provide well-being, enjoyable to receive and to practice.

This treatment is already offered to the patients at the ICO, in priority while the first course of chemotherapy, but in an informal way. I has been noticed a better-being after the TM, and an increase of demand from the patients. This is why it would be interested to measure the evolution of quality of life of those patients having a chemotherapy for a breast cancer getting or not a TM.

DETAILED DESCRIPTION:
The participation of the study will be offered to each patient coming for a first course of chemotherapy at the hospital day care for an adjuvant breast cancer. The tracking of the eligible patient will be done during the registration for the schedule.

The filling of the questionnaires will occur at the 4 first courses (C1 to C4). The Touch Massage will be offered for the 3 first courses of chemotherapy (C1 to C3). The patient can refuse the TM but she will have to fill the questionnaires.

At each moment, the patient can withdraw from the study, the TM can be offered according to the availability of the team and of the choice of the patient during the course of chemotherapy.

The questionnaire collection will be done in the patient's room. The quality of life will be evaluated based on the questionnaires EORTC, QLQ C30 and BR23 at C1 and C2. The evaluation of the quality of life at the fourth course will allow to estimate the quality of life after 3 complete courses of chemotherapy. Alongside, the anxiety will be evaluated with the anxiety scale STAI from C1 to C3, when the patient just arrives in the service and before she leaves. At the fourth course, the questionnaire will be filled only at the arrival.

After the filling of the questionnaires, the patient will be seen by the medical doctor of the service and the nurse who will take charge of her for the chemotherapy.

According the availability of the service, the patient will receive the TM if she wants. A member of the nursing staff formed to the TM (formation dispensed to the ICO) will perform the TM. It will be done during the chemotherapy, during the perfusion of ENDOXAN, which takes an hour. The TM will last 20 minutes. In this way, the TM will not delayed, prolonged and disturb the treatment. At C4, there will not be a TM.

ELIGIBILITY:
Inclusion Criteria:

* women between 18 and 70 years old
* patient with histologically confirmed breast cancer
* adjuvant situation
* spoken language : french
* patient who never had chemotherapy in the past

Exclusion Criteria:

* Patient unable to sit
* Malformation of the back
* Wound at the level of the zones to massage
* Patient placed under the authority of a tutor
* Pregnant patient

Ages: 18 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women between 18 and 70 years old with an adjuvant breast cancer histologically characterized
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2020-05-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the quality of life of patients with an adjuvant breast cancer treated at the ICO depending on the patient benefit or not from the TM during the chemotherapy in a hospital day care | 90 days
  Quality of life assessed using QLQ-C30 (Quality of Life of Cancer Patients) questionnaire. It is a general 30-item questionnaire composed by 5 functional scales, 3 symptom scales, a global health status and 5 single items assessing additional symptoms. The scales measures range score from 0 to 100. A high scale score represents a higher response level. For example, a high score for a functional scale represents a healthy level of functioning; a high score for the global health status represents a high quality of life; a high score for the symptom scales represents a high level of symptomatology or problems
Change from basline quality of life during breast cancer treatment | 90 days
  Quality of life assessed using BR23 questionnaire. It is a 23-item questionnaire to measure the functioning and the symptoms associated of breast cancer. The functional dimension is composed of several scales: the reflection of the body, sexual functioning, sexual pleasure and perspective of future. The symptom dimension is composed of different scales such as the systemic therapy, side effects, mammary symptoms, hand symptoms and hair loss.

SECONDARY OUTCOMES:
Estimate the prevalence of the patients interested by the TM as part of the adjuvant care of a breast cancer at the ICO site of Angers | 90 days
  The prevalence of the number of patients interested by the TM is the ratio between the patients responding "yes" to the question : "would you like to receive a Touch-Massage" and the number of patients included in the study.
Evaluate the benefits of the TM on the anxiety | 90 days
  Measure the anxiety with the help of the scale of the validated STAI (State Inventory Anxiety). A high score (more than 48 for men and 55 for women) represents a high level of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra PIQUIN, Nurse, Study Director — Insitut de Cancérologie de l'Ouest
Locations (1):
- Insitut de Cancérologie de l'Ouest, Angers, France

IPD SHARING:
Plan to Share IPD: No